CLINICAL TRIAL: NCT05394376
Title: DECIBEL(S): Determining Change In Blood Pressure Due to Environment and Loudness
Brief Title: Determining Change In Blood Pressure Due to Environment and Loudness
Acronym: DECIBEL(S)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Vital Strategies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: IRB00322730
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Environment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Inside private quiet1, Inside public loud, Inside public quiet, Inside private quiet2 (Other): The order of noise/environment for participants randomized to this arm will be:
  Inside private quiet1, Inside public loud, Inside public quiet, Inside private quiet2
  Interventions: Other: Level of noise and environment (public vs private) while taking blood pressure measurement
- Inside public loud, inside private quiet1, Inside public quiet, Inside private quiet2 (Other): The order of noise/environment for participants randomized to this arm will be:
  Inside public loud, inside private quiet1, Inside public quiet, Inside private quiet2
  Interventions: Other: Level of noise and environment (public vs private) while taking blood pressure measurement
- Inside public loud, inside public quiet, inside private quiet1, inside private quiet 2 (Other): The order of noise/environment for participants randomized to this arm will be:
  Inside public loud, inside public quiet, inside private quiet1, inside private quiet 2
  Interventions: Other: Level of noise and environment (public vs private) while taking blood pressure measurement
- Inside public quiet, inside public loud, inside private quiet1, inside private quiet2 (Other): The order of noise/environment for participants randomized to this arm will be:
  Inside public quiet, inside public loud, inside private quiet1, inside private quiet2
  Interventions: Other: Level of noise and environment (public vs private) while taking blood pressure measurement
- Inside public quiet, inside private quiet1, inside public loud, inside private quiet2 (Other): The order of noise/environment for participants randomized to this arm will be:
  Inside public quiet, inside private quiet1, inside public loud, inside private quiet2
  Interventions: Other: Level of noise and environment (public vs private) while taking blood pressure measurement
- Inside private quiet1, Inside public quiet, Inside public loud, inside private quiet2 (Other): The order of noise/environment for participants randomized to this arm will be:
  Inside private quiet1, Inside public quiet, Inside public loud, inside private quiet2
  Interventions: Other: Level of noise and environment (public vs private) while taking blood pressure measurement

INTERVENTIONS:
Other: Level of noise and environment (public vs private) while taking blood pressure measurement — Each participant will have 4 sets of 3 blood pressure measurements taken. The participants will be randomized to the order in which the level of noise in their environment changes and whether they are in a public or private setting prior to each set of measurements.

SUMMARY:
Determine the effects of environment and sound on initial and average triplicate screening blood pressure done according to clinical practice guidelines with an automated device.

Standardly obtained blood pressures obtained in a noisy, busy, public space will be higher than attended blood pressures obtained (1) in the same environment but with earplugs to minimize sound and (2) in a quiet, private space without surrounding activity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years

Exclusion Criteria:

* Hearing loss requiring hearing aids
* Presence of the following on both arms: rashes, gauze dressings, casts, edema, paralysis, tubes, open sores or wounds, A-V shunts.
* Being mentally impaired
* Being pregnant
* Arm circumference exceeding 55 cm.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Difference between first systolic BP and average of 3 systolic BPs from measurements (mmHg) | Time of reading up to 90 minutes
  Absolute difference between first systolic BP and average of 3 systolic BPs from measurements (mmHg) obtained in:
  * Inside public loud vs. Inside private quiet1
  * Inside public quiet vs. Inside private quiet1
  * Inside private quiet1 vs. Inside private quiet2
Difference between first diastolic BP and average of 3 diastolic BPs from measurements (mmHg) | Time of reading up to 90 minutes
  Absolute difference between (1) 1st diastolic BP and (2) average of 3 diastolic BP from measurements (mmHg) obtained with:
  * Inside public loud vs. Inside private quiet1
  * Inside public quiet vs. Inside private quiet1
  * Inside private quiet1 vs. Inside private quiet2
Systolic and Diastolic Differences in blood pressure measurement (mmHg) | Time of reading up to 90 minutes
  Systolic and Diastolic Difference of differences between:
  * (Inside private quiet 1 - Inside private quiet 2) and (Inside public loud- Inside private quiet 1)
  * (Inside private quiet1 - Inside private quiet2) and (Inside public quiet - Inside private quiet1)

SECONDARY OUTCOMES:
Difference in blood pressure measurement based on blood pressure level | Time of reading up to 90 minutes
  To determine the difference in blood pressure measurements based on blood pressure level (SBP ≥130 mmHg vs. SBP <130 mmHg)
Difference in blood pressure measurement based on age | Time of measurement up to 90 minutes
  To determine the blood pressure difference based on age (≥ 60 years vs. <60 years).
Difference in blood pressure measurement based on regular healthcare visits | Time of measurement up to 90 minutes
  To determine the blood pressure difference based on regular healthcare visits (>1 year vs. ≤ 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Brady, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Ishigami J, Liu H, Zhao D, Sabit A, Pathiravasan CH, Charleston J, Miller ER 3rd, Matsushita K, Appel LJ, Brady TM. Effects of Noise and Public Setting on Blood Pressure Readings : A Randomized Crossover Trial. Ann Intern Med. 2025 Feb;178(2):149-156. doi: 10.7326/ANNALS-24-00873. Epub 2025 Jan 28. PMID 39869911